CLINICAL TRIAL: NCT02206672
Title: EFFECTS OF THE MICRO REINJECTION OF AUTOLOGOUS ADIPOSE TISSUE IN THE FACE OF PATIENTS WITH SYSTEMIC SCLEROSIS
Acronym: FACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2014-A01014-43; 2014-12 (Other: AP HM)
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-09

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Micro reinjection of autologus adipose tissue (Other)
  Interventions: Other: Micro reinjection of autologus adipose tissue

INTERVENTIONS:
Other: Micro reinjection of autologus adipose tissue

SUMMARY:
This prospective single-center study evaluates a current care procedure. It includes 14 patients diagnosed with SSc according to the ACR/EULAR criteria or the Leroy & Medsger criteria of the disease. Patients are enrolled if they wish for a therapeutic care of their face, have a Mouth Handicap in Systemic Sclerosis (MHISS) score greater than 20 (scale 0-48), a modified Rodnan skin score upper or equal to 1 on the face (scale 0-3), and a mouth opening less than 55 millimeters. They should not have anticoagulant, anti-platelets aggregation medication or a daily steroid dose upper 20mg per day. Their BMI should exceed 17.

Micro fat grafting is a minimally invasive and usual procedure performed under local anesthesia. Fat tissue is harvested (around 50 milliliters) using a 14 gauge or 2 mm diameter cannula from areas around the knees, the abdomen or the hips under a gentle aspiration. Lipoaspirated fat is then filtrated by the PureGraft system that offers a sterile, closed, single-use system, leading to a fast, consistent and controlled preparation. Then, 10 to 25 milliliters of this purified fat product is transferred through a 21 gauge or 0.8 mm diameter cannula in two or four points of the face, with the entry points located around the mouth.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 or younger than 80 years.
* Suffering from systemic scleroderma.
* Patient follow-AP-HM.
* Score of 20 or greater MHISS.
* Score Rodnan level greater than or equal to one face.
* Mouth opening (inter-incisor distance) <5.5 cm
* Wishing to receive surgery at the face.

Exclusion Criteria:

* Less than 18 or greater than 80 age.
* Decaying history of abdominal surgery.
* Body mass index lower than 18.
* Coagulation disorders.
* Allergy to Xylocaine.
* Greater than 20mg / d steroids.
* Severe infection.
* Inmates.
* Pregnant women.
* Adults protected by law (under guardianship and trusteeship).
* No affiliation to a social security scheme.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
improvement of the MHISS score | 12 months
  The MHISS questionnaire is chosen as it specifically assesses disability involving the mouth and the face in SSc patients.

SECONDARY OUTCOMES:
evaluate the effect of the procedure on quality of life | 12 months
  Health Assessment Questionnaire adapted to scleroderma, SHAQ
evaluate the effect of the procedure on face pain | 12 months
  face pain scale (VAS 0-100)
evaluate the effect of the procedure on skin fibrosis | 12 months
  skin fibrosis is measured by Rodnan skin score for the face, mouth opening measure and cutometry)
evaluate the effect of the procedure on physical face changes | 12 months
  physical face changes is evaluated by standard and 3D photographs.

CONTACTS AND LOCATIONS:
Overall Officials: brigitte GRANEL, MD, Principal Investigator — AP HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France